CLINICAL TRIAL: NCT04367766
Title: Management of the Fresh Extraction Socket in the Aesthetic Area: Alveolar Ridge Preservation vs Immediate Implant Placement vs Delayed Implant Placement
Brief Title: Management of the Fresh Extraction Socket in the Aesthetic Area
Acronym: IIP/ARP/SH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Specialistico Odontoiatrico, Rome (Network)
Responsible Party: Principal Investigator, Marco Clementini, Research Fellow, Centro Specialistico Odontoiatrico, Rome
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIP/ARP/SH
Record Dates: First submitted 2020-04-25; First posted 2020-04-29 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Tooth Extraction Status Nos; Dental Implant; Bone Augmentation; Soft Tissue Augmentation
Keywords: Immediate implant placement; alveolar ridge preservation; delayed implant placement; PROMs; implant health; volumetric analysis; tissue augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Implant Placement (Active Comparator): prosthetically driven immediate implant placement (TLC implant, Straumann) with bone substitute (BioOss Collagen, Geistlich) filling the gap between the buccal socket wall and the implant surface and a collagen matrix (Fibrogide, Geistlich) positioning at the vestibular aspect to increase soft tissue volume, with immediate (non occlusal loading) prosthetic provisionalization.
  Interventions: Procedure: Prosthetically driven implant placement
- Alveolar Ridge Preservation (ARP) + Delayed Implant Placement: (Active Comparator): ARP performed with bone substitute (BioOss Collagen, Geistlich) and a collagen matrix placed to seal the socket entrance (Mucograft Seal, Geistlich). After 4 months of healing a prosthetically driven implant (TLC implant, Straumann) will be placed with adjunctive GBR procedure with bone substitute (BioOss Collagen, Geistlich) and a collagen membrane (BioGide, Geistlich) if buccal bone will be < 2 mm and soft tissue augmentation with a collagen matrix (Fibrogide, Geistlich) if soft tissue thickness will be < 2mm
  Interventions: Procedure: Prosthetically driven implant placement
- Spontaneous Healing + Delayed Implant Placement (Active Comparator): extraction socket will be left to heal spontaneously. After 4 months of healing a prosthetically driven implant (TLC implant, Straumann) will be placed with adjunctive GBR procedure with bone substitute (BioOss Collagen, Geistlich) and a collagen membrane (BioGide, Geistlich) if buccal bone will be < 2 mm, and soft tissue augmentation with a collagen matrix (Fibrogide, Geistlich) if soft tissue thickness will be < 2mm .
  Interventions: Procedure: Prosthetically driven implant placement

INTERVENTIONS:
Procedure: Prosthetically driven implant placement — Insertion of an osseointegrated implant into the bone of anterior maxilla/mandible, following the right prosthetic plan
  Other Names: Prosthetically driven implant installation

SUMMARY:
After atraumatic tooth extraction and the assessment of the feasibility of immediate implant placement, patients will be randomly assigned to one of three treatment concepts:

1. Immediate Implant Placement and Immediate Provisionalization
2. Alveolar Ridge Preservation. After 4 months of healing an implant will be placed with simultaneous GBR and/or Soft Tissue Augmentation procedures, if needed.
3. Spontaneous Healing of the socket. After 4 months of healing, an implant will be placedwith simultaneous GBR and/or Soft Tissue Augmentation procedures, if needed.

In all groups, four months after implant placement, a prosthesis will be delivered. From this experimental period onward, patients will be scheduled for maintenance. Clinical, radiographic and volumetric assessment will be performed by clinicians not involved in the surgery and blind with respect to treatment assignment at 1, 3 and 5 years post loading.

DETAILED DESCRIPTION:
The overall objective of this study will be to compare the three treatment modalities after tooth extraction (immediate implant placement, alveolar ridge preservation, spontaneous healing) in terms of:

* patient-related (morbidity) outcomes during surgical procedure and the first 2 weeks after the surgical procedure
* cost-effectiveness ratio (treatment time, number of surgeries, number of appointments and overall appointments time, need for bone and soft tissue augmentation, overall costs) at the time of prosthesis delivery
* volumetric bone and soft tissue changes of the site before treatment (prior to tooth extraction), 4 months after tooth extraction, 1, 3 and 5 years after final prosthesis.
* clinical, radiographic, aesthetic and patient-related (satisfaction) outcomes at the time of prosthesis delivery and 1, 3 and 5 years after final prosthesis.
* Implant Success and Survival at 1, 3 and 5 years after final prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* single tooth extraction in the anterior region of the dentition (including premolars) to be extracted
* smoking no more than 10 cigarettes/day,
* periodontal health (BoP < 10%) and good plaque control (< 20%)
* absence of symptomatic periapical radiolucencies, acute abscesses at the site of extraction,
* extraction sites with less than 30% loss of one or more walls
* adequate quantity and quality of native bone to achieve primary stability

Exclusion Criteria:

* growing patients
* patients with autoimmune disease, uncontrolled diabetes or immunocompromised
* history of head and neck radiation for cancer treatment,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of adjunctive bone and soft tissue augmentation procedures need. | during implant placement
  Number of participants with the need for adjunctive reconstructive hard tissue procedure during implant placement will be evaluated as a frequency (Yes/No) after a digital prosthetically driven implant placement. The need for soft tissue augmentation during implant placement will be evaluated as a frequency (Yes/No) by a blinded examiner in case of buccal soft tissue thickness < 2mm assessed at 3mm apical to the full thickness flap margin with a caliber.

SECONDARY OUTCOMES:
Peri-Implant Health | 1, 3, 5 years post loading
  Peri-implant health will be assessed as a frequency (Yes/No) at 1, 3, 5 years after prosthetic crown delivery by a blinded examiner in case of: absence of clinical signs of inflammation, absence of bleeding and/or suppuration on gentle probing, no increase in probing depth compared to previous examinations, absence of bone loss beyond crestal bone level changes resulting from initial bone remodeling

OTHER OUTCOMES:
Patient Reported Outcome Measurements | crown delivery, 1, 3, 5 years post loading
  Patient's satisfaction with the final result will be assessed by means of a 100 mm VAS scale ranging from 0 (no satisfaction) to 100 (best possible satisfaction), recording patient's experience
Clinical parameters: Probing Depth (PD) and Recession (REC) | crown delivery, 1, 3, 5 years post loading
  Probing Depth (PD) and Recession (REC) will be recorded in mm. with a periodontal probe (P-UNC 15, Hu Friedy) inserted with a standardised pressure into the peri-implant sulcus at 6 sites per implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual)
Clinical parameters: Bleeding on Probing (BoP) | crown delivery, 1, 3, 5 years post loading
  Bleeding on Probing (BoP) will be recorded as presence/absence with a periodontal probe (P-UNC 15, Hu Friedy) inserted with a standardised pressure into the peri-implant sulcus at 6 sites per implant (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual)
Marginal Bone Level (MBL) | crown delivery, 1, 3, 5 years post loading
  Marginal Bone Level (MBL) will be evaluated by a blinded examiner analysing an intra-oral radiograph on a computer software (Image J), as the distance in mm. between the smooth-rough interface and the mesial and distal bone level. The radiographs will be performed using a customized PVS bite block and an alignment device
Aesthetic | crown delivery, 1, 3, 5 years post loading
  Aesthetic will be evaluated by a blinded examiner analysing pictures using the modified pink and white aesthetic score (PES/WES system, Belser et al. 2009) and giving a score from 0 to 20.
Volumetric bone and soft tissue changes | before tooth extraction, 4 months after tooth extraction, at prosthetic crown delivery and 1, 3 and 5 year after crown delivery.
  Volumetric bone change will be assessed by a blinded examiner analysing on a computer software (SMOP) DICOM files from cone-beam computed tomography (CBCT) scan. Contour soft tissue change and buccal soft tissue volume will be assessed by a blinded examiner analysing on a computer software (SMOP) STL files from digital impression. Dynamic Soft tissue healing will be assessed by a blinded examiner analysing superimposition on a computer software (SMOP) of DICOM files (from CBCT) and STL files (from digital impression)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Clementini, DDS, PhD, Principal Investigator — Centro Specialistico Odontoiatrico, Rome
Locations (1):
- Centro Specialistico Odontoiatrico (CSO), Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results will be presented in open access publication in international peer-reviewed journal
Supporting Information: Study Protocol
Time Frame: From the publication acceptance by the international peer-reviewed journal
Access Criteria: Open access publication

REFERENCES:
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112
- [Background] Clementini M, Agostinelli A, Castelluzzo W, Cugnata F, Vignoletti F, De Sanctis M. The effect of immediate implant placement on alveolar ridge preservation compared to spontaneous healing after tooth extraction: Radiographic results of a randomized controlled clinical trial. J Clin Periodontol. 2019 Jul;46(7):776-786. doi: 10.1111/jcpe.13125. Epub 2019 May 31. PMID 31050359